CLINICAL TRIAL: NCT06816563
Title: Prediction of Version Outcomes for External Maneuvers of Breech Fetus by Assessment of Breech Progression Angle (breech Progression Angle)
Brief Title: Prediction of Version Outcomes for External Maneuvers of Breech Fetus by Assessment of Breech Progression Angle
Acronym: ECV
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ECV
Record Dates: First submitted 2024-12-30; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Breech Presentation
Keywords: Breech fetus
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Breech presentation complicates about 3-4% of single pregnancies at term. Although vaginal delivery is also possible in breech presentations, this is associated with an increased risk of fetal morbidity and mortality. The cephalic version for external maneuvers is an obstetric procedure that allows conversion of an abnormal presentation/situation (breech or transverse) to a cephalic presentation by applying pressure to the maternal abdomen. Over the years, many authors have analyzed numerous factors that might be associated with an increased likelihood of successful maneuvering. Over time, transperineal ultrasonography has proven to be a valid, objective, and highly reproducible tool for the assessment of fetal head progression during delivery in conjunction with examination. The Angle of Progression (AoP) is the angle between the line passing through the longitudinal axis of the pubic symphysis and the line passing through the inferior border of the pubic symphysis and tangent to the fetal skull. AoP is an accurate and reproducible parameter for the assessment of fetal head descent during labor, with a strong correlation with the mode of delivery. The investigators are not aware of any studies that have established the role of transperineal ultrasound in assessing podietal engagement and its role in predicting the success of the cephalic version maneuver, an aspect the investigators want to explore with this study.

DETAILED DESCRIPTION:
Patients will be recruited before starting the cephalic version for external maneuvers. An ultrasound evaluation will be performed for each patient before the external maneuver version of breech fetus; specifically, the following will be performed:

* Transabdominal ultrasound for evaluation of the following parameters: type of breech presentation, estimated fetal weight (according to Hadlock), maximum amniotic fluid flap, position of the placenta (anterior/posterior or fundic), angle between the fetal spine at the cervical level and the fetal occiput (occipital-spine angle).
* Transperineal ultrasound for evaluation of the following parameters: Breech Progression Angle (BPA), Subpubic Arch (SPA).

If the external maneuver version is successful, an additional transperineal ultrasound will be performed for evaluation of Angle of Progression (AoP).

After delivery, data will be recorded regarding mode of delivery, indication for operative delivery (in case of cesarean section or obstetric suction), neonatal arterial and venous pH, possible admission to the NICU. These data will be collected by consulting the medical records of recruited patients. The population will be recruited as part of the normal care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age with a single pregnancy at term (37-42 gestational weeks) with a fetus in breech presentation
* Acquisition of Informed Consent Form

Exclusion Criteria:

* Oligohydramnios: maximum flap < 2cm
* Placenta previa
* Uterine malformations
* Regular uterine dynamics
* Metrorrhagia
* Contraindications to vaginal delivery
* Premature rupture of membranes
* Nonreassuring cardiotocographic tracing
* Previous uterine surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with a single full-term pregnancy (37-42 gestational weeks) with a fetus in breech presentation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of new ultrasound indexes (Breech Progression Angle, BPA) | During the ultrasound performed before the version for external maneuvers of breech fetus
  Evaluation using transperineal ultrasonography, the role of a new ultrasound index (Breech Progression Angle, BPA) in predicting the success of external maneuver version of breech fetus

CONTACTS AND LOCATIONS:
Overall Officials: Aly Mohamed Alaaeldin Kamaleldin Aly Youssef, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna